CLINICAL TRIAL: NCT02994485
Title: Evaluation Of The Portal Pressure By Doppler Ultrasound In Cirrhotic Patients Before And After Simvastatin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sherief Abd-Elsalam, Principle investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Nadia Elwan
Record Dates: First submitted 2016-12-13; First posted 2016-12-15 (Estimated); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Portal Hypertension
MeSH Terms: conditions — Hypertension, Portal | interventions — Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Simvastatin (Active Comparator): Simvastatin 20 mg/day for two weeks (increased to 40 mg/day at day 15) for another two weeks
  Interventions: Drug: Simvastatin
- no treatment (No Intervention): no treatment

INTERVENTIONS:
Drug: Simvastatin — Simvastatin 20 mg/day for two weeks (increased to 40 mg/day at day 15) for another two weeks plus the routine treatment
  Other Names: Corvast
  Arms: Simvastatin

SUMMARY:
Portal hypertension is not a disease in itself. Rather, it is an indication of an illness, caused mostly by chronic lesions of the liver because of distinct causes, such as viral infection, chronic alcoholism, or metabolic disorders. Other reasons include splanchnic vascular diseases (for example, obstruction of the portal or the hepatic veins). Portal hypertension is defined as a pressure in the portal vein exceeding the vena cava pressure by more than 5 mm Hg.

DETAILED DESCRIPTION:
Indeed, use of simvastatin might attenuate liver fibrosis in patients with chronic C infection, it may also reduce hepatic vascular resistance and portal pressure by improving liver generation of nitric oxide and hepatic endothelial dysfunction in patients with cirrhosis, so it could be an effective therapy for portal hypertension. It might even improve survival of patients with cirrhosis after variceal bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Positive diagnosis of cirrhosis by US (coarse echogenic pattern, bulky caudate lobe, attenuated hepatic veins)
* Clinical manifestations of portal hypertension (as esophageal varices ,splenomegaly, ascites and encephalopathy grade I-II)

Exclusion Criteria:

* Pregnancy
* Hepatic encephalopathy grade III-IV
* Hepatocellular carcinoma
* Treatment with statins in the previous 3 months
* Hypersensitivity to statins
* Previous surgical shunt or TIPS
* Treatment with calcium channel blockers

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-10; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Number of Patients with Reduced Portal Pressure After Intervention | 6 Months
  the number of Patients with Reduced Portal Pressure After Intervention

CONTACTS AND LOCATIONS:
Overall Officials: NADIA ELWAN, PROFESSOR, Principal Investigator — Tanta university hospital; RAAFAT SALAH, PROFESSOR, Study Chair — Tanta university hospital; MANAL HAMISA, Ass Prof, Study Chair — Tanta university hospital; EBTESAM A SHADY, BACHELOR, Study Chair — Tanta University hospital
Locations (1):
- Sherief Abd-Elsalam, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Elwan N, Salah R, Hamisa M, Shady E, Hawash N, Abd-Elsalam S. Evaluation of portal pressure by doppler ultrasound in patients with cirrhosis before and after simvastatin administration - a randomized controlled trial. F1000Res. 2018 Mar 1;7:256. doi: 10.12688/f1000research.13915.1. eCollection 2018. PMID 29707200